CLINICAL TRIAL: NCT02152852
Title: Peer Support for Achieving Independence in Diabetes (Peer AID)
Brief Title: Peer Support for Achieving Independence in Diabetes
Acronym: Peer-AID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Public Health - Seattle and King County (Other Government)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 5R18DK088072 (NIH); 5R18DK088072 (NIH)
Record Dates: First submitted 2014-05-23; First posted 2014-06-02 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Community Health Worker Intervention (Experimental): Community Health Worker Intervention-home visits from community health workers providing education and support for self-management of type 2 diabetes, resources for diabetes control, and assistance in effective communication with medical providers
  Interventions: Behavioral: Community Health Worker Intervention
- Usual Care Control Group (No Intervention): Usual Care Control Group- Usual care is defined as services received by participants in the absence of the intervention plus information about community resources that support diabetes self-management (such as classes and support groups) and educational pamphlets.

INTERVENTIONS:
Behavioral: Community Health Worker Intervention — For the intervention group, a trained Community Health Worker (CHW) will provide education, support and service coordination through in-home visits. The CHW will first make an in-home assessment visit. At the assessment visit, the participant has the opportunity to ask questions and sign written consent. During this visit, the CHW assesses the participant's history with diabetes, medication adherence, self-management activities, healthcare utilization and will administer a finger stick blood test for HbA1c and a full lipid panel. After enrollment, the participant receives up to five follow-up educational visits 0.5, 1.5, 3.5, 7 and 10 months later. In addition to scheduled visits, the CHWs work with their participants on an as-needed basis via telephone, or additional home visits.
  Arms: Community Health Worker Intervention

SUMMARY:
The purpose of this study is to test the hypotheses that CHWs providing in-home support for self-management of type 2 diabetes, resources for diabetes, and assistance in effective linkage and communication with medical providers will: (1) improve HbA1c (primary outcome) and secondary outcomes including lipids, blood pressure, health care utilization, and health-related quality of life; (2) improve diabetes self-management, including self-efficacy, physical activity, nutrition, and medication adherence; and (3) be cost-effective and feasible.

DETAILED DESCRIPTION:
The investigators will implement a randomized trial that will enroll 286 participants, from three different sites, to compare a CHW intervention consisting of home visits, telephone support, and linkage to appropriate community-based group activities compared to usual care. Usual care is defined as the medical care received by participants in the absence of the intervention plus information about community resources that support diabetes self-management (such as classes and support groups) plus educational pamphlets. The investigators will randomize an equal number of participants to the intervention and control groups.

After collecting baseline data, we will assign participants to study groups using a stratified, permuted block design with varying block size. The investigators will stratify by site to ensure an approximately equal number of treatment and control subjects at each site and also meet the site-specific recruitment targets. The nature of the intervention makes it impossible to blind participants and staff to group assignment.

CHWs will primarily work with participants in their homes, and will also link them to community resources that support self-management. CHWs will make up to 5 home visits for each participant in the intervention arm. To assure that the program is feasible to implement in a variety of clinical settings, to assure external validity of the study, and to assess potential for adoption, the CHWs will be based at the local public health department and participants will be recruited from a county hospital system, a community clinic and a Veteran Affairs (VA) hospital.

Specific aims of the proposal are to examine the effect of the intervention on physiologic markers of disease control (HbA1c, lipids, blood pressure), participant self-efficacy, self-management behaviors quality of life and utilization and costs. The investigators will measure other demographic, medical and psychosocial patient level characteristics that could potentially modify the effects of the intervention. At the end of the study period, CHWs will visit usual care participants so that they receive many of the potential benefits received by intervention group members.

The investigators will use mixed methods to assess translation of the research models into practice.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes and HbA1c of 8.0% or greater
* Household income less than 250% of the federal poverty level
* Residence within target area of King County, Washington
* Age 30-70 years.
* Primary language spoken by participant is English or Spanish

Exclusion Criteria:

* Type 1 diabetes
* Pregnant
* Unable to provide informed consent
* End-stage renal disease (ESRD), dementia, or a terminal illness
* Plans to move within the next two years or is homeless
* Other mental or physical disability making it impossible to participate in the protocols

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2011-11; Primary Completion 2015-04 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Improvement in HbA1c | One Year
  HbA1c will be assessed at baseline and then again at 12 months.

SECONDARY OUTCOMES:
Improvement in lipids | One Year
  Lipids will be assessed at baseline and again at 12 months.
Improvement in blood pressure | One Year
  Will assess blood pressure at baseline and 12 months.
Healthcare Utilization | One Year
  Will assess healthcare utilization at baseline and at 12 months.
Physical and mental functioning | One year
  The project will assess changes in physical and mental functioning at baseline and again at 12 months. The measure used will be the Short Form (SF)-12, a 12-question survey that asks participants to recall their physical and mental status over a four week time frame. Changes measured include: role limitations caused by physical health, emotional problems, physical functioning, and general health over a four week period.

CONTACTS AND LOCATIONS:
Overall Officials: Karin Nelson, MD, MSHS, Principal Investigator — VA Puget Sound; James Krieger, MD, MPH, Principal Investigator — Public Health Seattle King County